CLINICAL TRIAL: NCT03650205
Title: Ivabradine to Prevent Anthracycline-induced Cardiotoxicity: a Randomized Clinical Trial
Brief Title: Ivabradine to Prevent Anthracycline-induced Cardiotoxicity
Acronym: IPAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar, Clinical director of the Instituto do Coracao, Faculdade de Medicina, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 42559415520020065
Record Dates: First submitted 2018-08-13; First posted 2018-08-28 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Neoplasms; Heart Failure; Cardiotoxicity; Chemotherapy Effect; Oncology
MeSH Terms: conditions — Neoplasms; Heart Failure; Cardiotoxicity | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivabradine (Active Comparator): Patients will receive ivabradine just before anthracycline chemotherapy, 5 mg per oral twice daily, until one month after the last chemotherapy session.
  Interventions: Drug: Ivabradine
- Placebo (Placebo Comparator): Patients will receive placebo just before anthracycline chemotherapy, one capsule per oral twice daily, until one month after the last chemotherapy session.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — Ivabradine capsule
  Arms: Ivabradine
Drug: Placebo — Placebo oral capsule.
  Other Names: Placebo oral capsule
  Arms: Placebo

SUMMARY:
Anthracyclines are associated with cardiotoxic effects. Previous studies suggest that enalapril, and or carvedilol, protect against cardiovascular effects of these drugs.

Ivabradine selectively reduces heart rate through inhibition of the cardiac pace maker IF channel, thus prolonging the duration of spontaneous depolarization in the sinus node. Additionally, ivabradine might preserve myocardial perfusion without negative inotropic effect and probably maintain cardiac contractility despite the reduction of heart rate.

Ivabradine has been shown to improve outcome in patients with heart failure and angina. The aim of this study is to evaluate whether ivabradine might prevent anthracycline-induced cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-year-old or older;
* Cancer diagnosis;
* Chemotherapy with anthracycline;
* Written informed consent

Exclusion Criteria:

* Chronic Kidney Disease (Creatinine clearance inferior to 30mL/min/1.73m2)
* Bradycardia (heart rate less than 60 beats per minute)
* Atrial fibrilation;
* Previous diagnosis of heart failure;
* Pregnancy;
* History of previous hypersensibility to the study drug;
* Participating in another study protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Ventricular function | 365 days after randomization
  Reduction in global longitudinal strain of at least 10% (GLS)

SECONDARY OUTCOMES:
Composite endpoint of mortality or major cardiovascular outcomes | 365 days after randomization
  Composite endpoint of mortality or major cardiovascular outcomes (defined as acute myocardial infarction, heart failure, inappropriate sinus tachycardia and arrhythmia)
Left ventricular dysfunction | 365 days after randomization
  Incidence of left ventricular (LV) dysfunction defined as reduction of LV ejection fraction by 10%.
Incidence of myocardial injury | 90 days after randomization
  Levels of NT-proBNP and high-sensitivity cardiac troponin T
Incidence of myocardial injury | 180 days after randomization
  Levels of NT-proBNP and high-sensitivity cardiac troponin T
Incidence of myocardial injury | 365 days after randomization
  Levels of NT-proBNP and high-sensitivity cardiac troponin T
Diastolic dysfunction | 365 days after randomization
  Assessment by echocardiography the incidence of diastolic dysfunction using the following parameters: peak E-wave velocity, peak A-wave velocity, mitral valve (MV) E/A ratio, MV deceleration time, pulsed-wave tissue doppler imaging e' velocity, Mitral E/e', left atrium maximum volume index, pulmonary vein(PV) systole(S) wave, PV diastole (D) wave, continuous wave (CW) doppler: tricuspid regurgitation, systolic jet velocity; Color M- mode.
Ventricular function | 180 days after randomization
  Reduction in global longitudinal strain of at least 10% (GLS)

OTHER OUTCOMES:
Composite endpoint of mortality or major cardiovascular outcomes | yearly after randomization until 5 years
  Composite endpoint of mortality or major cardiovascular outcomes (defined as acute myocardial infarction, heart failure, inappropriate sinus tachycardia and arrhythmia)
Left ventricular dysfunction | 180 days after randomization
  Incidence of left ventricular (LV) dysfunction defined as reduction of LV
Incidence of myocardial injury | 90 days after randomization
  Levels of NT-proBNP and high-sensitivity cardiac troponin T
Incidence of myocardial injury | 180 days after randomization
  Levels of NT-proBNP and high-sensitivity cardiac troponin T
Diastolic dysfunction | 180 days after randomization
  Assessment by echocardiography the incidence of diastolic dysfunction using the following parameters: peak E-wave velocity, peak A-wave velocity, mitral valve (MV) E/A ratio, MV deceleration time, pulsed-wave tissue doppler imaging e' velocity, Mitral E/e', left atrium maximum volume index, pulmonary vein(PV) systole(S) wave, PV diastole (D) wave, continuous wave (CW) doppler: tricuspid regurgitation, systolic jet velocity; Color M- mode.
Adverse events | 180 days after randomization
  bradycardia, hypertension, atrial fibrillation, luminous phenomena, syncope, hypotension, erythema, rash, diplopia, vertigo, urticaria
Adverse events | 365 days after randomization
  bradycardia, hypertension, atrial fibrillation, luminous phenomena, syncope, hypotension, erythema, rash, diplopia, vertigo, urticaria
Heart rate variability | 180 days after randomization
  Assessment of heart variability through 24-hour holter the following parameters: mRR - ms, SDNN - ms, SDANN - ms, SDNNi - ms, rMSSD-ms, NN50, pNN50.
Oxygen consumption (VO2) | 180 days after randomization
  Measurement of VO2 by cardiopulmonary exercise test
Ventilatory equivalents for oxygen (VE/VO2) and for carbon dioxide (VE/VCO2) | 180 days after randomization
  Measurement of ventilatory equivalents for oxygen (VE/VO2) and for carbon dioxide (VE/VCO2) by cardiopulmonary exercise test
Left Ventricular Dimensions | yearly after randomization until 5 years
  LV diastolic diameter, LV diastolic diameter, LV diastolic diameter
Left ventricular geometry and mass | yearly after randomization until 5 years
  LV mass, Septal thickness, Posterior wall thickness
Subgroup analyses regarding the primary outcome | 365 days after randomization
  Type of cancer, gender, age

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizk SI, Costa IBSDS, Cruz CBBV, Pileggi B, de Almeida Andrade FT, Gonzalez TB, Bittar CS, Fukushima JT, Quintao VC, Osawa EA, Alves JBS, Fonseca SMR, Garcia DR, Pereira J, Buccheri V, Avila J, Kawahara LT, Barros CCS, Ikeoka LT, Nakada LN, Fellini M, Rocha VG, Rego EM, Hoff PMG, Filho RK, Landoni G, Hajjar LA. Randomized, Placebo-Controlled, Triple-Blind Clinical Trial of Ivabradine for the Prevention of Cardiac Dysfunction During Anthracycline-Based Cancer Therapy. J Am Heart Assoc. 2025 May 20;14(10):e039745. doi: 10.1161/JAHA.124.039745. Epub 2025 May 13. PMID 40357644